CLINICAL TRIAL: NCT04109768
Title: Culinary Medicine Intervention to Empower Pre-Adolescent Children to Help Their Families to Improve Nutrition Literacy, Self-Image and Well-Being
Brief Title: Hands On Nutrition Education to Improve Childhood Health
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left university
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Krista Casazza, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 300002498
Record Dates: First submitted 2019-09-25; First posted 2019-09-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Health Behavior; Nutrition Poor
MeSH Terms: conditions — Health Behavior; Malnutrition | interventions — Nutritional Status; Exercise

STUDY DESIGN:
Intervention Model Description: pre post intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hands on Nutrition Education (Experimental): Nutrition and activity intervention to improve behaviors pre to post
  Interventions: Behavioral: nutrition and activity

INTERVENTIONS:
Behavioral: nutrition and activity — 16 sessions; nutrition 8; activity 8- 45 minutes to improve health and nutrition literacy

SUMMARY:
The main goals of this study is to better understand how an experiential cooking, movement and mindfulness intervention influence elementary school children at Spring Valley School. program diet, fitness, metabolic outcomes, health literacy and overall well-being. Specifically, the role of the novel empowering experiential learning through a cooking and fitness intervention activities will play on health literacy and metabolic outcomes, engagement in fitness and motivation, and stress levels will be evaluated.

DETAILED DESCRIPTION:
Nutrition and mindful movement program activities will take place during the school day. Children will be given the opportunity understand the value of quality nutrition in the prevention com-morbidities of treatment and poor lifestyle choices. The intervention will consist of ten sessions. This includes pre- and post-assessments (weeks 1 and 10) and eight weekly 1-hour interactive culinary medicine education sessions. Children will be asked questions about their diet, feelings, physical activity. Height, weight, waist circumference, and grip strength will also be measured. This will take about one hour prior to beginning the education portion of our program. Each week, \a nutrition lecture, a cooking demo and fitness activities will be completed over two-45 minutes sessions during PE class. These hands-on applied nutrition sessions include fundamental of nutrition, cooking skills, cooking skills, and activities. Experiential or hands-on applied learning, including culturally appropriate meal preparation and personalized nutrition and mindful movements, represents a potential tool to increase adolescent health literacy as well as empower adolescent to engage their families. Cooking as medicine helps people make the healthy behavior changes they are seeking because it allows hands-on teaching and learning in a fun interactive environment, without stigma. This strategy encompasses combination of thinking and doing skills that are applied during home food preparation, as well as conceptual and perceptual abilities on food handling, safety and storage, and other factors related to nutrition. The delivery of cooking as medicine programs serves as a way to improve and promote confidence, well-being, and enhance meal quality and preparation practices and offer a valuable platform to engage children and families via inclusive social activities, whilst positively impacting their dietary profiles and health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* speak and read English able to ambulate student at selected school

Exclusion Criteria:

* medical condition precluding participation

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
health literacy | 10 weeks
  A questionnaire to evaluate pre and post health literacy specific to nutrition will be used
metabolic outcome | 10 weeks
  glucose, insulin, lipid profile will be evaluated by biochemical analysis following a blood draw
self-efficacy | 10-weeks
  A self-efficacy questionnaire evaluating child's perceived capacity to prepare and consume healthy meals will be assessed.

IPD SHARING:
Plan to Share IPD: No